CLINICAL TRIAL: NCT06766968
Title: Prolonged Compression Therapy Following Foam Sclerotherapy of Varicose Veins
Brief Title: Prolonged Compression Following Foam Sclerotherapy
Acronym: ProCOMFFS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Kirill Lobastov, Professor, Pirogov Russian National Research Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ProCOMFFS
Record Dates: First submitted 2025-01-04; First posted 2025-01-09 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Chronic Venous Disorder; Varicose Veins Leg
Keywords: varicose veins; chronic venous disease; sclerotherapy; medical compression stockings
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Intervention Model Description: A single-center, open, superiority randomized controlled trial with a blinded outcome assessor.
Who Masked: Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: MCS for 1 month (Experimental): The patient will be prescribed to use medical compression stockings (MCS of class 2 of "RAL GZ 387" standard with a pressure of 23-32 mm Hf at the ankle) continuously for 7 days between the sessions and after the last session of foam-form sclerotherapy. After that, he should continue wearing the MCS during the day (put it on within 30 minutes after getting out of bed, remove it within 30 minutes before going to sleep, and wear it for at least 12 hours a day) for 28 days.
  Interventions: Device: Graduated Compression Stocking: 1 month using
- Group 2: MCS for 1 week (Active Comparator): The patient will be prescribed to use medical compression stockings (MCS of class 2 of "RAL GZ 387" standard with a pressure of 23-32 mm Hf at the ankle) continuously for 7 days between the sessions and after the last session of foam-form sclerotherapy. After that he will stop using MCS.
  Interventions: Device: Graduated Compression Stocking: 1 week using

INTERVENTIONS:
Device: Graduated Compression Stocking: 1 month using — Class 2 (RAL-GZ 387 standard: 23-32 mm Hg at the ankle level) above-knee graduated compression stockings
  Arms: Group 1: MCS for 1 month
Device: Graduated Compression Stocking: 1 week using — Class 2 (RAL-GZ 387 standard: 23-32 mm Hg at the ankle level) above-knee graduated compression stockings
  Arms: Group 2: MCS for 1 week

SUMMARY:
Foam-form sclerotherapy is an effective method for eliminating varicose veins, which can be used alone or in combination with other interventions (laser or radiofrequency ablation, cyanoacrylate glue embolization) in the treatment of chronic venous disease of the lower limbs. Sclerotherapy is utilized to address both primary and recurrent varicose veins, and it is associated with a low rate of complications. Among the adverse effects, the most common is skin hyperpigmentation (darkening of the skin with the formation of stripes of shades of brown directly above the treated veins), with an occurrence rate reaching 6-53% within the first month following the procedure. Still, it resolves independently in 70% of cases within 6 months. An essential component of sclerotherapy is compression therapy through bandages or medical stockings, which helps accelerate the absorption of veins and improve the aesthetic results of treatment. Meanwhile, the optimal duration for wearing compression stockings after performing foam-form sclerotherapy of varicose tributaries has not been established.

DETAILED DESCRIPTION:
Foam-form sclerotherapy effectively eliminates varicose veins, which can be used independently or combined with trunkal ablation to treat chronic venous disease. Sclerotherapy eliminates both primary and recurrent varicosity and is associated with a low frequency of complications. Among the adverse events, the most common is skin hyperpigmentation, with a 6-53% detection rate during the first month after the procedure. However, it resolves spontaneously in 70% of cases within a follow-up period of up to 6 months. Compression therapy is currently considered a mandatory component of sclerotherapy for telangiectasias and reticular veins. Studies indicate that its use for periods ranging from 3 days to 4 months can reduce the incidence of hyperpigmentation by 1.5 to 5 times.

Meanwhile, the role of elastic compression during foam-from sclerotherapy of varicose tributaries has not yet been fully clarified. According to a recent randomized controlled study CONFETTI, wearing medical compression stockings (MCS) with a pressure of 18-24 mm Hg at the ankle continuously for 7 days compared to applying a compression bandage for 24 hours was associated with a reduction in pain intensity. Still, it did not affect the severity of chronic venous disease, quality of life, time to return to normal activity, technical success of the procedure, or the frequency of bruising. However, the risk and severity of hyperpigmentation and other adverse effects were not investigated. Therefore, there is a need to determine the feasibility of prolonged use of MCS after foam-form sclerotherapy for varicose veins.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Varicose veins of the lower extremities of clinical class C2 according to CEAP (Clinical, Etiological, Anatomical, Pathophysiological) classification;
* Scheduled foam-form sclerotherapy of varicose tributaries as an independent intervention or after trunkal ablation;
* Absence of initial skin pigmentation, including that associated with previously performed trunk ablation;
* Absence of indications for long-term use of compression therapy, including the clinical class of chronic venous disease C3-C6 and persistence of vein-specific symptoms;
* Signed informed consent to participate in the study.

Exclusion Criteria:

* History of deep vein thrombosis;
* Contraindications or restrictions to foam-form sclerotherapy;
* Contraindications or restrictions to long-term use of compression therapy;
* Inability or difficulty in independently putting on MCS;
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with hyperpigmentation at 28 days | 28 days
  Assessed by a blinded expert based on the analysis of photographic images of the legs in 4 projections (front, back, right, and left) as the presence of a linear area of skin in various shades of brown in the projection of sclerosed veins.

SECONDARY OUTCOMES:
Intensity of the hyperpigmentation at 28 days | 28 days
  Assessed by a blinded expert based on the analysis of photographic images of the legs in four projections (front, back, right, and left) using a 4-level Likert's-like scale: 0 - no pigmentation, 1 - mild hyperpigmentation, 2 - moderate hyperpigmentation, 3 - severe hyperpigmentation.
Number of patients with hyperpigmentation at 6 months | 6 months
  Assessed by a blinded expert based on the analysis of photographic images of the legs in 4 projections (front, back, right, and left) as the presence of a linear area of skin in various shades of brown in the projection of sclerosed veins.
Intensity of hyperpigmentation at 6 months | 6 months
  Assessed by a blinded expert based on the analysis of photographic images of the legs in four projections (front, back, right, and left) using a 4-level Likert's-like scale: 0 - no pigmentation, 1 - mild hyperpigmentation, 2 - moderate hyperpigmentation, 3 - severe hyperpigmentation.
Intensity of spontaneous pain in the sclerosed vein at 28 days | 28 days
  The intensity of pain over the sclerosed vein is assessed subjectively by the patient on a 10-cm numeric rating scale at rest. Ranges from 0 (no pain) to 10 (pain of the maximal intensity).
Intensity of spontaneous pain in the sclerosed vein at 6 months | 6 months
  The intensity of pain over the sclerosed vein is assessed subjectively by the patient on a 10-cm numeric rating scale at rest. Ranges from 0 (no pain) to 10 (pain of the maximal intensity).
Intensity of stimulated pain in the sclerosed vein at 28 days | 28 days
  The intensity of pain over the sclerosed vein is assessed subjectively by the patient on a 10-cm numeric rating scale during compression of the vein. Ranges from 0 (no pain) to 10 (pain of the maximal intensity).
Intensity of stimulated pain in the sclerosed vein at 6 months | 6 months
  The intensity of pain over the sclerosed vein is assessed subjectively by the patient on a 10-cm numeric rating scale during compression of the vein. Ranges from 0 (no pain) to 10 (pain of the maximal intensity).
Number of patients with resorption of sclerosed veins at 6 months | 6 months
  The absence of any signs of previously obliterated veins (visible veins, thickened areas) upon examination and palpation by the Investigator.
The value of VCSS at 28 days | 28 days
  The severity of chronic venous disease (CVD) in the target lower limb is assessed during clinical examination using the updated Venous Clinical Severity Score (VCSS). Ranges from 0 to 30. The maximal score indicates more severe CVD.
The value of VCSS at 6 months | 6 months
  The severity of chronic venous disease (CVD) in the target lower limb is assessed during clinical examination using the updated Venous Clinical Severity Score (VCSS). Ranges from 0 to 30. The maximal score indicates more severe CVD.
The value of CIVIQ-20 score at 28 days | 28 days
  The quality of life is assessed by the patient independently according to the vein-specific questionnaire Chronic Lower Limb Venous Insufficiency Questionnaire - 20 items (CIVIQ-20). range 0-100, a minimal score indicates the best quality of life.
The value of CIVIQ-20 score at 6 months | 6 months
  The quality of life is assessed by the patient independently according to the vein-specific questionnaire Chronic Lower Limb Venous Insufficiency Questionnaire - 20 items (CIVIQ-20). range 0-100, a minimal score indicates the best quality of life.
Level of comfort with the use of MCS at 7 days | 7 days
  The patients subjectively assess their comfort when using MCS using a 10-cm numeric rating scale, which ranges from 0 (no comfort) to 10 (absolute comfort).
Level of comfort with the use of MCS at 28 days | 28 days
  The patients of Group 1 (Experimental) subjectively assess their comfort when using MCS using a 10-cm numeric rating scale, which ranges from 0 (no comfort) to 10 (absolute comfort).
Compliance with the use of MCS | 28 days
  Compliance with the use of MCS is assessed based on the study of the patient's diaries in Group 1 (Experimental) as a proportion of the number of days when the patient used MCS for at least 12 hours to the total duration of prescribed compression (28 days) represented as a percentage (n[MCS]/28*100%). It ranges from 0% (no compliance) to 100% (absolute compliance).
Difference in the interface pressure below the MCS | 28 days
  The level of interface pressure under the MCS is measured in real-time using the "PicoPress" manometer ("Microlab", Italy) at points B (ankle), B1 (midway between B and C), C (widest part of the calf), D (head of the fibula), F (mid-thigh), and G (upper third of the thigh) in mm Hg. The measurements are performed in Group 1 (Experimental) at the randomization before the first application of the stocking (day 0) and on day 28. The difference is reported as the pressure at the B1 point on day 0 minus pressure at the B1 point on day 28 (pressure B1[d0] - pressure B1[d28]. It may range in a broad spectrum of numbers from 0 (no changes in the pressure over time) to minus figures (pressure increases over time) or plus figures (pressure decreases over time). It is assumed that the range should be between -10 and +10 mm Hg.
Number of patients with symptomatic venous thromboembolism | 6 months
  Symptomatic venous thromboembolism includes deep vein thrombosis, pulmonary embolism, and superficial vein thrombosis of the vein not previously treated with foam-form sclerotherapy confirmed by appropriate medical imaging (duplex ultrasound, CT-pulmonary angiography).
Number of patients with phlebitis of the sclerosed vein | 6 months
  Phlebitis of a sclerosed vein refers to the appearance of signs of inflammation (hyperemia, swelling, pain) in the projection of a previously treated with foam sclerotherapy vein.
Number of patients with skin lesions | 6 months
  Skin lesions related to the use of MCS refer to the emergence of dryness, peeling, rashes, hyperemia, swelling, weeping, and breaches in skin integrity while wearing compression stockings.
Number of patients with adverse events | 6 months
  Refers to any other adverse events despite skin lesions that could be associated with using MCS of foaf-form sclerotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Kirill Lobastov, PhD, Principal Investigator — Pirogov Russian National Research Medical University
Locations (1):
- MedSwiss Private Clinic, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
By the personal request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After results publication indefinitely
Access Criteria: By the personal request